CLINICAL TRIAL: NCT05000359
Title: A Mobile Phone Intervention to Promote Adherence to Survivorship Care Among Adolescent and Young Adult Cancer Survivors
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-000440
Record Dates: First submitted 2021-07-09; First posted 2021-08-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Survivors of Childhood Cancer

STUDY DESIGN:
Intervention Model Description: Ten AYA survivors will be recruited to participate in the expanded 12-week text messaging intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA Text messaging intervention (Other): Ten AYA survivors will be recruited to participate in the expanded 12-week text messaging intervention.
  Interventions: Behavioral: text messaging intervention

INTERVENTIONS:
Behavioral: text messaging intervention — Ten AYA survivors will be recruited to participate in the expanded 12-week text messaging intervention.

SUMMARY:
Adolescents and young adults (AYA) survivors of childhood cancer receive inadequate surveillance for treatment-related late effects. This study evaluates the acceptability and feasibility of a mobile phone messaging intervention targeting behavior changes related to receiving survivorship care among AYA survivors.

Content from an existing text-messaging survivorship education intervention will be adapted to a novel text-messaging platform, Chorus. Ten AYA survivors will be recruited to participate in the expanded 12-week text messaging intervention. In-depth interviews will be conducted with each participant during the study, and a focus group with all participants will be conducted at the end of the study. Qualitative analysis will determine areas for improvement in the text messaging intervention in order to ensure acceptability and feasibility in AYA survivors. The text messaging intervention on Chorus will be adapted to better suit the needs of AYA survivors based on the results of the qualitative analysis. Mobile phone interventions offer a cost-effective, age-appropriate approach to AYA survivorship care education. If effective, the text-messaging intervention will be evaluated in a randomized, controlled pilot trial to improve rates of survivorship care and clinical outcomes for AYA survivors.

DETAILED DESCRIPTION:
Aim 1: To adapt and enhance an existing text messaging intervention to an expanded two-way multi-media mobile phone messaging platform (Chorus) that will improve knowledge regarding the risk of late effects among AYA survivors, intent to seek recommended survivorship care, and completion of standard survivorship care goals. a. both two-way text messaging to improve Children?s Oncology Group (COG) survivorship guideline adherence b. web-based educational content for survivors of key survivorship messages regarding risk for late effects and need for ongoing survivorship care c. Monthly peer navigation phone calls to address barriers and promote retention d. utilization of pre and post-test questionnaires for participants to access and complete within the Chorus platform Aim 2: To test the acceptability and feasibility of the expanded mobile phone intervention content to improve messaging and strategies for survivorship care using qualitative methodologies and applying the Technology Acceptance Model (TAM) within a sample of AYA survivors. a. perceived usefulness of the text messaging system b. perceived ease of use of the text messaging system c. effect of the text messaging system on health-related behavior intent

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 to 39 years at the time of enrollment
* Patient must reside in the greater Los Angeles area.
* Patients must have received survivorship care at the University of California at Los Angeles (UCLA)
* Patients must be fluent in English.
* Patients must be off cancer therapy for at least one year.
* Patients must have personal access to a smart phone with text messaging and internet and/or data capability.

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Mobil Phone Muti-Media messaging | one month
  Acceptability and feasibility of an expanded mobile phone intervention as assessed by key informant interview questions and a focus group discussion developed based on the Technology Acceptance Model: (a) perceived usefulness of the text messaging system for completing ASAP goals, (b) perceived ease of use of the text messaging system for completing ASAP goals, and (c) effect of the text messaging system on intent to complete ASAP goals. The assessment will be qualitative only.
  The Technology Acceptance Model (TAM) evaluates how likely a user of new technology will accept and continue to use the new technology. TAM posits that if the technology is perceived as useful, easy to use, and increases intent to use - then the technology is more likely to be accepted. Interview questions and focus group discussion points will ask about these criteria. If responses satisfy the TAM criteria, this supports mobile phone intervention as acceptable and feasible for use in AYA cancer survivors.

SECONDARY OUTCOMES:
Key Informant Interview regarding risk for late effects due to prior cancer treatment and intent to seek survivorship care. | up to 1 year
  Themes for refinement of the text messaging intervention as assessed by key informant interview questions designed to elicit feedback on features of the mobile phone intervention that could improve knowledge regarding risk for late effects and intent to seek survivorship care.
  Hypothetical example: Collectively, participants believed that the intervention's incorporation of weblinks and phone numbers to community resources clarified their risk for late effects as a cancer survivor.
Key Informant Interview to identify themes from which the mobile phone intervention will be refined in order to improve its potential impact on the completion of participants' Adolescent and Young Adult Survivorship Action Plan (ASAP) goals. | up to 1 year
  Key informant interviews with YA survivors regarding their experience during the mobile phone intervention will identify themes from which the mobile phone intervention will be refined in order to improve its potential impact on the completion of participants' Adolescent and Young Adult Survivorship Action Plan (ASAP) goals.
  Theoretical example: Collectively, participants believed the appointment reminders provided by the mobile phone intervention made it more likely for them to attend their survivorship care clinic appointment and, thus, complete their ASAP goal (adherence to survivorship care).

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Garcia, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No